CLINICAL TRIAL: NCT05164861
Title: Assessment of Safety and Efficacy of Non-alcoholic Pasteurized Beverage Based on Kombucha, Enriched With Inulin and Vitamins in Patients With Constipations
Brief Title: Safety and Efficacy of Non-alcoholic Beverage Based on Kombucha in Patients With Constipations
Acronym: Kombucha
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vasily Isakov (Other)
Collaborators: Azbuka vkusa (Unknown); Russian Science Foundation (Other); Federal Research Centre of Nutrition, Biotechnology and Food Safety (Unknown)
Responsible Party: Sponsor-Investigator, Vasily Isakov, Professor, MD, PhD, AGAF, Russian Academy of Medical Sciences
Organization: Russian Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-76-30014/2021K-OGIG
Record Dates: First submitted 2021-12-04; First posted 2021-12-21 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Irritable Bowel Syndrome With Constipation; Constipation-predominant Irritable Bowel Syndrome
Keywords: specialized food product; kombucha; safety; efficacy; constipation; functional food
MeSH Terms: conditions — Constipation | interventions — Inulin; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/kombucha-based beverage (Experimental): Subjects randomized to this group will receive newly developed food product - non-alcoholic pasteurized beverage based on kombucha enriched with inulin and vitamins, flavoured as "Black currant with juniper" or "Strawberries with lime" or 'Mango with passion fruit"
  Interventions: Dietary Supplement: kombucha-based beverage
- Control (No Intervention): Subjects of this group will receive standard diet with similar quantity of water as in experimental group

INTERVENTIONS:
Dietary Supplement: kombucha-based beverage — kombucha-based beverage: drinking water, black tea, kombucha, inulin, vitamins (B1, B2, B6, niacin, folic acid). Nutritional value in 100 ml: carbohydrates - 2.57 g (including sucrose - 0.22 g, glucose - 1.32 g, fructose - 1.03 g), inulin - 1.15 g (46%*), vitamin B1 - 0.4 mg (29%*), B2 - 0.21 mg (13%*), B6 - 0.48 mg (24%*), niacin - 2.74 mg (15%*), folic acid - 24.0 mcg (12%*). Energy value/Caloric content - 54 kilojoules/13 kcal (* - % of the recommended daily allowance, according to the Technical regulations of the Customs Union #022/2011). Flavours, identical by nutrient's content and nutrients density: black currant berries & juniper berries, or strawberries & lime leaves, or passion fruit & mango.
  Portion's volume - 220 ml. Daily intake: 1 portion
  Other Names: Kombucha enriched with inulin, vitamins and flavours
  Arms: Intervention/kombucha-based beverage

SUMMARY:
Single centre, open-label, non-randomized study is planned to proof the concept of safety and efficacy of newly developed specialized food product - non-alcoholic pasteurized beverage based on kombucha, enriched with inulin and vitamins in patients with constipations

DETAILED DESCRIPTION:
This single-center open-label non-randomized study is planned to proof the concept on safety and efficacy of newly developed specialized food product - non-alcoholic pasteurized beverage based on kombucha, enriched with inulin and vitamins in patients with irritable bowel syndrome with constipations.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate (based on signed informed consent form)
* irritable bowel syndrome with predominant constipation, per Rome IV criteria (Recurrent abdominal pain on average at least 1 day/week in the last 3 months, associated with two or more of the following criteria: related to defecation; associated with a change in frequency of stool; associated with a change in form (appearance) of stool - Bristol stool scale types 1 or 2. Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis),

Exclusion Criteria:

* pregnant or breast-feeding women;
* intolerance of kombucha or any component of the product;
* history of abdominal surgery;
* the use of concomitant medications able to affect bowel motility;
* general condition of a patient making the appropriateness of his participation in the study questionable;
* chronic decompensated disorders of any organs and systems;
* mean daily caloric intake less than 800 kcal and more than 6000 kcal
* inability to follow standard iso-caloric diet and standard volume of water consumption (1.5-2 litres a day)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Change of number bowel movements | two weeks
  Number of bowel movements per week will be assessed per patients self report
Change of stool type | a week
  Stool type assessed per the Bristol stool scale (from type 1 to type 7; where type 1 - separate hard lumps, like nuts, type 7 - watery, no solid pieces, entirely liquid stool - diarrhoea)

SECONDARY OUTCOMES:
Adverse events | two weeks
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, Professor, Principal Investigator — Federal Research Center of Nutrition and Biotechnology
Locations (1):
- Gastroenterology and Hepatology, FRC Nutrition and Biotechnology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Blinded to personal data individual participant data may be shared per reasonable request after study completion
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: study data will available during 5 years after study completion
Access Criteria: per reasonable request to principal investigator
URL: https://grant.rscf.ru/

REFERENCES:
- [Derived] Isakov VA, Pilipenko VI, Vlasova AV, Kochetkova AA. Evaluation of the Efficacy of Kombucha-Based Drink Enriched with Inulin and Vitamins for the Management of Constipation-Predominant Irritable Bowel Syndrome in Females: A Randomized Pilot Study. Curr Dev Nutr. 2023 Nov 24;7(12):102037. doi: 10.1016/j.cdnut.2023.102037. eCollection 2023 Dec. PMID 38149073
- [Derived] Pilipenko VI, Isakov VA, Morozov SV, Vlasova AV, Kochetkova AA. [Efficacy of newly developed kombucha-based specialized food product for treatment of constipation-predominant irritable bowel syndrome]. Vopr Pitan. 2022;91(5):95-104. doi: 10.33029/0042-8833-2022-91-5-95-104. Epub 2022 Aug 30. Russian. PMID 36394933
- See also: Rome IV criteria — https://theromefoundation.org/rome-iv/rome-iv-criteria/